CLINICAL TRIAL: NCT05033496
Title: The Yield of Postnatal Thyroid Function Test in Term Newborn Infants in the Well Baby Nursery in Addition to the National Screening Test Program
Brief Title: The Yield of Postnatal Thyroid Function Test in the Well Baby Nursery
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Neonatologist, Hillel Yaffe Medical Center
Other Study IDs: 0128-21-HYMC-IL
Record Dates: First submitted 2021-08-25; First posted 2021-09-02 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroid Function Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn infants: Newborn infants born in our medical center
  Interventions: Diagnostic Test: Thyroid function test

INTERVENTIONS:
Diagnostic Test: Thyroid function test — Thyroid function test

SUMMARY:
Thyroid function test are performed in the well baby nursery to newborn infants of mothers with hypothyroidism, or as part of neonatal jaundice investigation. As thyroid function test are also part of the national screening test program, the investigators raised the option that the above management is unnecessary, and managed a study to investigate it.

DETAILED DESCRIPTION:
Thyroid function test are performed in the well baby nursery to newborn infants of mothers with hypothyroidism, or as part of neonatal jaundice investigation. As thyroid function test are also part of the national screening test program, the investigators raised the option that the above management is unnecessary, and managed a study to investigate it.

The study is retrospective. About 4000 infants are born in the center every year. The investigators wish to examine data for 10 years, i.e. about 40000 files.

The investigators will collect all the national screening test program results and compare them to the thyroid function test performed in that center.

ELIGIBILITY:
Inclusion Criteria:

* Infants born in our medical center
* Term infants
* Admitted to well baby nursery and stayed there until discharge

Exclusion Criteria:

* Preterm infants
* Transferred to neonatal intensive care unit for any reason

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants born in our medical center
Sampling Method: Non-Probability Sample
Enrollment: 40601 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Hypothyroidism found in local test was missing by national screening test | 10 years
  The proportion of missed hypothyroidism in screening test (missing = found in local test and missed in national screening test)
Hypothyroidism found in screening test was missing in local test | 10 years
  The proportion of missed hypothyroidism in local test (missing = found in national screening test and missed in local test)

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be erased.

REFERENCES:
- [Background] van Trotsenburg P, Stoupa A, Leger J, Rohrer T, Peters C, Fugazzola L, Cassio A, Heinrichs C, Beauloye V, Pohlenz J, Rodien P, Coutant R, Szinnai G, Murray P, Bartes B, Luton D, Salerno M, de Sanctis L, Vigone M, Krude H, Persani L, Polak M. Congenital Hypothyroidism: A 2020-2021 Consensus Guidelines Update-An ENDO-European Reference Network Initiative Endorsed by the European Society for Pediatric Endocrinology and the European Society for Endocrinology. Thyroid. 2021 Mar;31(3):387-419. doi: 10.1089/thy.2020.0333. PMID 33272083
- [Background] Alexander EK, Pearce EN, Brent GA, Brown RS, Chen H, Dosiou C, Grobman WA, Laurberg P, Lazarus JH, Mandel SJ, Peeters RP, Sullivan S. 2017 Guidelines of the American Thyroid Association for the Diagnosis and Management of Thyroid Disease During Pregnancy and the Postpartum. Thyroid. 2017 Mar;27(3):315-389. doi: 10.1089/thy.2016.0457. PMID 28056690
- [Background] American Academy of Pediatrics; Rose SR; Section on Endocrinology and Committee on Genetics, American Thyroid Association; Brown RS; Public Health Committee, Lawson Wilkins Pediatric Endocrine Society; Foley T, Kaplowitz PB, Kaye CI, Sundararajan S, Varma SK. Update of newborn screening and therapy for congenital hypothyroidism. Pediatrics. 2006 Jun;117(6):2290-303. doi: 10.1542/peds.2006-0915. PMID 16740880